CLINICAL TRIAL: NCT05313542
Title: Effect of Physical Activity in the Format of Self-defence Training for Depressive Symptoms - A Pilot Randomised Controlled Trial
Brief Title: Physical Activity in the Format of Self-defence Training for Depressive Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY021
Record Dates: First submitted 2022-03-29; First posted 2022-04-06 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Depressive Symptoms
Keywords: Self Defence Training; Physical Activity
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity Group (PA group) (Experimental): The PA group will receive a 6-week home-based self-defence training programme consisting of 120 min video training (including daily practice time) per week. Self-report questionnaires will be collected at baseline, immediate post-intervention, and 4-week follow up assessments.
  Interventions: Behavioral: Physical Activity
- Waitlist Group (WL group) (Other): The waitlist group will receive access to the programme at the end of study.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Physical Activity in the format of Self-defence Training

SUMMARY:
Inadequate mental health care capacity is a long-standing issue in Hong Kong (Yang & Mak, 2020). For example, a recent study predicts an additional 12% service need for specialist psychiatric care (Ni et al., 2020). It would be helpful to develop interventions that would ease the high demand of the health care system. Physical activity has been shown to reduce depressive symptoms in a number of studies (Bellón et al., 2021; Josefsson et al., 2014; Kvam et al., 2018; Schuch et al., 2016). Its flexibility and low-cost nature make physical activity a good intervention option for depressed individuals to do it anytime and anywhere.

This study aims to investigate the effect of physical activity intervention in the format of self-defence training on depressive symptoms. Around 40 eligible participants with at least moderate level of depressive symptoms will be randomly assigned to the physical activity (PA) group and waitlist (WL) control group. The PA group will receive a 6-week home-based self-defence training programme consisting of 120 min video training (including daily practice time) per week. Self-report questionnaires will be collected at baseline, immediate post-intervention, and 4-week follow up assessments. The primary outcome measure will be the Patient Health Questionnaire-9 to evaluate depression severity. Secondary outcomes will include psychological health symptoms, sleep quality, lifestyle, and quality of life. This research will provide new perspectives on the application of physical activity in the form of self-defence training as an intervention for depressive individuals.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 65 years old
* Hong Kong Residents
* Patient Health Questionnaire (PHQ-9) score ≥ 10; and
* Willingness to provide informed consent and comply with the trial protocol.

Exclusion Criteria:

* Patients with any cardiovascular diseases
* Receiving psychological treatment or medication for psychiatric disorders
* Participated in self defence training in the past 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Patient Health Questionnaire (PHQ-9) | Baseline, immediately post-intervention, 4-week follow-up
  The PHQ-9, a 20-item questionnaire used for screening, diagnosing, monitoring and measuring the severity of depression, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day).

SECONDARY OUTCOMES:
Change in the Short Form (Six-Dimension) Health Survey (SF-6D) | Baseline, immediately post-intervention, 4-week follow-up
  SF-6D is a preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.
Change in the International Physical Activities Questionnaire - Chinese version (IPAQ-C) | Baseline, immediately post-intervention, 4-week follow-up
  Participants' sitting time, walking time and moderate and vigorous physical activity are assessed by 5 questions from the short form of the International Physical Activity Questionnaire - Chinese version. Participants' engagement in brief strength and stamina-enhancing activity were assessed by asking the number of days they engaged in physical activity while seated and standing in the last seven days.
Change in the Insomnia Severity Index (ISI) | Baseline, immediately post-intervention, 4-week follow-up
  The ISI is a 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.
Change in Hospital Anxiety and Depression Scale (HADS-14) | Baseline, immediately post-intervention, 4-week follow-up
  HADS is a 14-item self-rated questionnaire which consists of two 7-item subscales that measure the presence of anxiety and depression symptoms respectively. Each item is rated on a 4-point-scale (0-3) by the participant. The greater the score, the more psychologically distressed the respondent is.
Change in Multidimensional Fatigue Inventory (MFI-20) | Baseline, immediately post-intervention, 4-week follow-up
  The MFI-20 assesses the severity of fatigue covering the following dimensions: general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.
Change in Credibility-Expectancy Questionnaire (CEQ) | Baseline, immediately post-intervention, 4-week follow-up
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.
Change in Treatment Adherence Survey (TAS) | Baseline, immediately post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided